CLINICAL TRIAL: NCT03277690
Title: A Double-blind, Placebo-Controlled, Randomized Withdrawal Following Open Label Therapy Study to Assess the Safety and Efficacy of Levoketoconazole (2S, 4R-ketoconazole) in the Treatment of Endogenous Cushing's Syndrome
Brief Title: A Study to Assess the Safety and Efficacy of Levoketoconazole in the Treatment of Endogenous Cushing's Syndrome.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cortendo AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COR-2017-01
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Endogenous Cushing's Syndrome
Keywords: Cushing Syndrome, Adrenocortical Hyperfunction
MeSH Terms: conditions — Cushing Syndrome; Adrenocortical Hyperfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Levoketoconazole (Experimental): Double blind withdrawal phase: Levoketoconazole (up to a dose of 1200 mg); Double blind restoration phase: Levoketoconazole plus Placebo
  Interventions: Drug: Levoketoconazole
- Placebo (Placebo Comparator): Double blind withdrawal phase: Placebo; Double blind restoration phase: Placebo plus Levoketoconazole
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levoketoconazole — During the double-blind Withdrawal Phase, patients will receive up to 1200 mg levoketoconazole daily.
  During the double-blind Restoration Phase, patients will receive levoketoconazole plus placebo.
  Other Names: COR-003
  Arms: Levoketoconazole
Drug: Placebo — During the double-blind Withdrawal Phase, patients will receive placebo tablets.
  During the double-blind Restoration Phase, patients will receive placebo plus levoketoconazole.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled withdrawal and rescue/restoration study in subjects with endogenous Cushing's Syndrome (CS) previously treated with single-arm, open-label levoketoconazole that will assess efficacy, safety, tolerability, and pharmacokinetics of levoketoconazole.

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo-controlled withdrawal and rescue/restoration study in subjects with endogenous CS that will assess efficacy, safety, tolerability, and Pharmacokinetics (PK) of levoketoconazole. There are two populations (cohorts) of subjects: (1) subjects which were previous levoketoconazole study completers and (2) subjects that are levoketoconazole treatment naïve subjects.

Study methodology varies by cohort prior to randomization only. Following initial screening (washout as needed) and Dose Titration and Maintenance Periods, as applicable, this study will be conducted in two double-blind phases (a Withdrawal Phase and a Restoration Phase). The levoketoconazole-naïve cohort will need to go through the Dose Titration and Maintenance Phase. The longest anticipated total study participation duration is approximately 51 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

SONICS STUDY COMPLETERS:

Completed the final SONICS visit (M12) and have demonstrated maintenance of clinical response on a stable Therapeutic Dose of levoketoconazole for at least 12 weeks prior to study entry.

ALL OTHERS:

* Confirmed newly diagnosed, persistent or recurrent endogenous Cushing's syndrome of any etiology, except secondary to malignancy (including pituitary or adrenal carcinoma).
* Elevated mean 24-hour Urinary Free Cortisol (UFC) levels at least 1.5X upper limit of the normative range of the study's central laboratory assay and from a minimum of three measurements from adequately collected urine.
* Presence of abnormal values from at least one of these two diagnostic tests:

  * Abnormal Dexamethasone Suppression Test (DST) OR
  * Elevated late night salivary cortisol concentrations (at least two measurements) each greater than the upper limit of the study's central laboratory normative range
* Non-candidates for CS-specific surgery, refuse surgery or surgery will be delayed until after study completion and agree to complete this study prior to surgery.
* If post-surgical for CS-specific surgery, then no significant post-operative sequelae remain and the risk of such sequelae is considered negligible.

EXCLUSION CRITERIA:

Subjects will be excluded from the study if ANY of the following criteria are met (NOTE: exclusion criteria apply to and must be assessed in both cohorts):

* Enrolled in SONICS but have not completed SONICS through Visit M12.
* Pseudo-Cushing's syndrome based on assessment of the Investigator.
* Cyclic Cushing's syndrome with multi-week periods of apparent spontaneous CS remission.
* Non-endogenous source of hypercortisolism, including pharmacological corticosteroids or ACTH.
* Radiotherapy of any modality directed against the source of hypercortisolism within the last 5 years.
* Treatment with mitotane within 6 months of enrollment.
* History of malignancy, including adrenal or pituitary carcinomas (other than low-risk, well-differentiated carcinomas of thyroid, breast or prostate that are very unlikely to require further treatment in the opinion of the treating physician, or squamous cell or basal cell carcinoma of the skin).
* Clinical or radiological signs of compression of the optic chiasm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Valencia, MD, Study Director — Cortendo AB
Locations (45):
- United States (13):
  - Keck Medical Center University of Southern California HCII, Internal Medicine - Keck Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Cedars-Sinai Pituitary Center, Los Angeles, California
  - UCLA School of Medicine, Medicine/Endocrinology Department, Los Angeles, California
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Emory University, Neurosurgery, Atlanta, Georgia
  - Northwestern University, Medicine - Endocrinology, Chicago, Illinois
  - Johns Hopkins University, Endocrinology Department, Baltimore, Maryland
  - University of Michigan, Comprehensive Endocrine Research, Internal Medicine - MEND, Ann Arbor, Michigan
  - Washington University School of Medicine, Endocrinology, St Louis, Missouri
  - Columbia University, College of P&S Medicine/Neuro-endocrine Unit, New York, New York
  - Memorial Sloan Kettering Cancer Center, Endocrinology, New York, New York
  - Oregon Health & Science University, Neurological Surgery, Portland, Oregon
  - Allegheny Neuroendocrinology Center, West Penn Allegheny Health System, Pittsburgh, Pennsylvania
- Bulgaria (3):
  - Alexandovska University Hospital, Clinic of Endocrinology & Metabolic Diseases, Sofia
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska" EAD Clinic of Endocrinology and Metabolic Diseases, Sofia
  - University Specialized Hospital for Active Treatment in Endocrinology (USHATE) I Klinika, Sofia
- Rigshospitalet, Copenhagen University Hospital, Endocrinology Department, Copenhagen, Denmark
- APHM Hôpital de la Conception, Service d'Endocrinologie, Diabète et Maladies Métaboliques, Marseille, Cedex 5, France
- Greece (5):
  - Evangelismos Athens General Hospital, Department of Endocrinology, Athens
  - General Hospital of Athens 'G. Gennimatas', Department of Endocrinology-Diabetes Centre, Athens
  - General Hospital of Athens 'Laiko', "National and Kapodistrian University of Athens Medical School Pathophysiology - Endocrinology", Athens
  - University General Hospital of Ioannina, Department of Endocrinology, Ioannina
  - Hippokration General Hospital, "Endocrinology and Diabetes Department, Thessaloniki
- Semmelweis Egyetem II. Belgyógyászati Klinika A.épület I.emelet ODM-labor, Budapest, Hungary
- Israel (3):
  - Bnai Zion Medical Center, Institute of Endocrinology, Haifa
  - Rabin Medical Center- Beilinson Hospital, "Institute of Endocrinology & Metabolism, Beilinson Campus", Petah Tikva
  - Tel-Aviv Sourasky Medical Center Institute of Endocrinology, Metabolism and Hypertension, Tel Aviv
- Italy (7):
  - Clinica di Endocrinologia e malattie del Metabolismo, Dipartimento Specialità Mediche, Ancona
  - University of Genova, Department of Internal Medicine & Medical Specialties (DiMI), Genova
  - AOU Policlinico G. Martino Sezione di Endocrinologia, Messina
  - AOU Federico II, Sezione di Endocrinologia (Edificio 1, Secondo Piano), Napoli
  - Policlinico Agostino Gemelli, Università Cattolica del Sacro Cuore, Endocrinology, Roma
  - Policlinico Universitario Sant'Andrea, Scienze Mediche, Roma
  - AOU Citta della Salure e della Scienza SC Endocrinologia, Diabetologia e Metabolismo, Torino
- Netherlands (2):
  - Leiden University, Leiden University Medical Center, Department of Endocrinology, Leiden
  - Erasmus Medical Center, Department of Internal Medicine, Rotterdam
- Poland (3):
  - Maria Sklodowska-Curie Memorial Institute - Cancer Center Gliwice Branch, Nuclear Medicine and Endocrine Oncology Department, Gliwice
  - Instytut Centrum Zdrowia Matki Polki, Oddział Endokrynologii i Chorób Metabolicznych, Lodz
  - Wojskowy Instytut Medyczny, Klinika Gastroenterologii, Endokrynologii I Chorob Wewnetrznych, Warsaw
- Romania (4):
  - Spitalul Clinic Judetean Mures, Compartimentul de Endocrinologie, Târgu Mureş, Mureș County
  - Spitalul Clinic Judetean de Urgenta "Pius Brinzeu", Departamentul de Endocrinologie, Timișoara, Timiș County
  - Institutul National de Endocrinologie C.I. Parhon, Sectia Clinica de Endocrinologie II, Patologia tiroidei de corelatie, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Sectia Clinica Endocrinologie, Cluj-Napoca
- Spain (2):
  - Hospital Universidad De La Ribera, Endocrinologia, Alzira, Valencia
  - Hospital Universitario Ramón y Cajal, Endocrinology and Nutrition, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Variable therapeutic response results in customized therapeutic doses (TD). The study design included an initial Titration-maintenance phase to identify a TD for each subject. It included a requirement for maintenance at TD for at least 4 weeks prior to entering the Randomized-withdrawal (RW) phase. Then a 1:1 RW to placebo was used to establish efficacy of the active therapy. 5 additional subjects began directly in RW after completing the parent study without requiring re-titration to TD.
Groups:
- Levoketoconazole: Double blind withdrawal phase: Levoketoconazole (up to a dose of 1200 mg); Double blind restoration phase: Levoketoconazole plus Placebo
  Levoketoconazole: During the double-blind Withdrawal Phase, patients will receive up to 1200 mg levoketoconazole daily.
  During the double-blind Restoration Phase, patients will receive levoketoconazole plus placebo.
- Placebo: Double blind withdrawal phase: Placebo; Double blind restoration phase: Placebo plus Levoketoconazole
  Placebo: During the double-blind Withdrawal Phase, patients will receive placebo tablets.
  During the double-blind Restoration Phase, patients will receive placebo plus levoketoconazole.
Period: Dose Titration and Maintenance
Arm/Group | Levoketoconazole | Placebo
Started | 79 | 0
Completed | 39 | 0
Not Completed | 40 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Sponsor decision - Randomization closed | 4 | 0
Not completed — Lack of Efficacy | 9 | 0
Not completed — Adverse Event | 15 | 0
Not completed — Withdrawal by Subject | 8 | 0
Period: Randomized Withdrawal
Arm/Group | Levoketoconazole | Placebo
Started (The number of participants starting this Period is not equal to the number who completed previous Period as 5 additional participants from the parent (SONICS) study directly entered the randomized withdrawal phase.) | 22 | 22
Subjects Which Were Previous Levoketoconazole Study Completers | 1 | 4
Subjects That Are Levoketoconazole Treatment naïve Subjects | 21 | 18
Completed | 21 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Restoration
Arm/Group | Levoketoconazole | Placebo
Started | 21 | 22
Subjects Which Were Previous Levoketoconazole Study Completers | 1 | 4
Subjects That Are Levoketoconazole Treatment naïve Subjects | 20 | 18
Completed | 21 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levoketoconazole | Placebo | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (11.97) | 43.6 (10.96) | 44.3 (11.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 34
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 20 | 22 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 18 | 22 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Greece | 4 | 0 | 4
  Netherlands | 0 | 1 | 1
  Romania | 1 | 3 | 4
  Hungary | 1 | 1 | 2
  United States | 3 | 5 | 8
  Poland | 1 | 1 | 2
  Italy | 3 | 4 | 7
  Israel | 1 | 3 | 4
  Bulgaria | 4 | 4 | 8
  France | 2 | 0 | 2
  Spain | 2 | 0 | 2
Receiving Anti-hypertensive Medication at Baseline [Count of Participants; unit: Participants]
  Yes | 16 | 14 | 30
  No | 6 | 8 | 14
Receiving Anti-diabetic Medication at Baseline [Count of Participants; unit: Participants]
  Yes | 8 | 6 | 14
  No | 14 | 16 | 30
Anatomical etiology of endogenous Cushing's syndrome [Count of Participants; unit: Participants]
  Cushing's Disease | 18 | 20 | 38
  Ectopic ACTH Secretion | 0 | 0 | 0
  Adrenal-Dependent | 3 | 1 | 4
  Unknown | 1 | 1 | 2
Mean Urinary Free Cortisol (mUFC) [Mean (Standard Deviation); unit: nmol/24 hours] | 738.69 (1067.025) | 411.59 (436.176) | 575.14 (822.384)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Loss of Therapeutic Response to Levoketoconazole Upon Withdrawing to Placebo Compared With the Proportion of Subjects With Loss of Therapeutic Response Upon Continuing Treatment With Levoketoconazole.
Description: Urinary free cortisol (UFC) level measurement: Loss of therapeutic response is inferred based on mUFC from three 24-hour UFC measurements obtained at any visit from second through final Randomized Withdrawal Phase visits (RW1 through RW5 inclusive) when: (1) mUFC is above 1.5X the ULN of the central laboratory's reference range, OR (2) mUFC is more than 40% above the baseline (RW0) value, if the RW0 value is above the ULN (i.e. >1.0X ULN)1, OR (3) an early rescue criterion is met.
Time Frame: max. 9.5 weeks
Population: Intent to Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Levoketoconazole | Placebo
Number analyzed (Participants) | 22 | 22
Participants | 9 | 21

ADVERSE EVENTS:
Time Frame: The intent to treat (ITT) population adverse events (AEs) are reported for the length of time the subject was in the randomized withdrawal (RW) phase, up to 9.5 weeks. The safety population AEs are reported for the full study length from informed consent to end of study, up to approximately 51 weeks.
Description: Untoward medical occurrence in a study subject that is temporally associated with the use of a medicinal product, regardless of its potential relationship to the medicinal product. An AE, therefore, can be any unfavorable or unintended sign, including an abnormal laboratory finding, symptom, or disease (new or exacerbated), whether related to the study drug or study conduct or not. NOTE: Abnormal values that reflect hypercortisolism (UFCs, LNSC and serum cortisol) will not be recorded as AEs.
Groups:
- Levoketoconazole-ITT RW Phase: During the double-blind Withdrawal Phase, patients will receive up to 1200 mg levoketoconazole daily.
- Placebo- ITT RW Phase: During the double-blind Withdrawal Phase, patients will receive placebo tablets.
- Safety Population: The safety population for the study overall (i.e., all phases combined), referred to all subjects who received at least 1 dose of study drug during any of the 3 study phases. This includes the subjects in the TM phase as well as the additional subjects who began directly in RW who completed the parent study and did not require re-titration to a therapeutic dose.
Arm/Group | Levoketoconazole-ITT RW Phase | Placebo- ITT RW Phase | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/84
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/22 | 13/84
Other Adverse Events (participants affected / at risk) | 11/22 | 10/22 | 73/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Levoketoconazole-ITT RW Phase (N=22) | Placebo- ITT RW Phase (N=22) | Safety Population (N=84)
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 2
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Levoketoconazole-ITT RW Phase (N=22) | Placebo- ITT RW Phase (N=22) | Safety Population (N=84)
Nausea (Gastrointestinal disorders) | 2 | 1 | 24
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 5
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 12
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 9
Fatigue (General disorders) | 2 | 1 | 10
Asthenia (General disorders) | 0 | 1 | 5
Oedema peripheral (General disorders) | 0 | 1 | 6
Pyrexia (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 10
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 21
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 19
Dizziness (Nervous system disorders) | 0 | 2 | 11
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood insulin increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Cortisol free urine increased (Investigations) | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 1 | 20
Insomnia (Psychiatric disorders) | 0 | 2 | 5
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 8
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 8
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 5
Nocturia (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 12
Lip Dry (Gastrointestinal disorders) | 0 | 0 | 8
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 4
Nasopharyngitis (Infections and infestations) | 0 | 0 | 7
Hypotension (Vascular disorders) | 0 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/90/NCT03277690/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT03277690/SAP_001.pdf